CLINICAL TRIAL: NCT04830735
Title: A Phase II Randomized Double-Blind Trial of Dasatinib Modulation of Hyperinflammation in Moderate and Severe Patients With COVID-19
Brief Title: Dasatinib for the Treatment of Moderate and Severe COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decided not to pursue study
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0S-20-5; NCI-2020-04367 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-20-5 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Symptomatic COVID-19 Infection Laboratory-Confirmed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (dasatinib anhydrous) (Experimental): Patients receive dasatinib anhydrous PO QD for 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib Anhydrous
- Arm II (placebo administration) (Placebo Comparator): Patients receive placebo PO QD for 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo Administration

INTERVENTIONS:
Drug: Dasatinib Anhydrous — Given PO
  Arms: Arm I (dasatinib anhydrous)
Drug: Placebo Administration — Given PO
  Arms: Arm II (placebo administration)

SUMMARY:
This phase II trial investigates how well dasatinib works in treating patients with moderate and severe COVID-19. Dasatinib is a drug used to treat chronic leukemia which may help reduce the strong inflammation caused by COVID-19 that can damage the lungs or other organs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients requiring intubation/ventilator support, requiring rescue with tocilizumab, or dying.

II. To determine 1 month survival.

SECONDARY OBJECTIVES:

I. To estimate the safety and tolerability of dasatinib anhydrous (dasatinib) in the setting of COVID-19 infection.

II. To determine change in C-reactive protein (CRP) levels after starting therapy.

III. To document activity of dasatinib in lessening cytokine release syndrome (CRS) and sequential organ failure assessment (SOFA) score.

EXPLORATORY OBJECTIVES:

I. Interleukin-6 /cytokine assay weekly on treatment protocol. II. Ferritin levels at study entry and every (q) 2 days on treatment protocol. III. D-dimer levels at study entry and q 2 days on treatment protocol.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive dasatinib anhydrous orally (PO) once daily (QD) for 14 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO QD for 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have laboratory test proven COVID19 and symptomatic disease requiring hospitalization: virological diagnosis of Sars-CoV2 infection (polymerase chain reaction [PCR]) within 14 days
* Able to sign informed consent for participation in the study
* Subject is hospitalized with one or more of the following:

  * Moderate disease: peripheral capillary oxygen saturation (SpO2) >= 93% on room air with one of the following risk factors for developing severe disease: age >= 60 years, history of hypertension, diabetes mellitus, cardiac disease, chronic lung disease, obesity (calculated body mass index [BMI] >= 30 kg/m^2), and cardiovascular disease, clinical and/or radiological evidence of chest involvement, CRP > 2X upper limit of normal, doubling of CRP in 24 hours where chest findings and CRP elevation not explained by other underlying disease.

After the first interim analysis, we may allow enrollment of severe disease COVID infected patients if safety and efficacy analysis appears favorable:

* Severe disease:

  * Respiratory rate >= 30 breaths/ minute (min)
  * SpO2 < 93% while breathing room air
  * Partial pressure of oxygen measurement (PaO2)/fraction of inspired oxygen (FiO2) =< 300 mmHg

    * Absolute neutrophil count (ANC) > 1000 (baseline blood counts)
    * Platelets > 50,000 / mmc (baseline blood counts)
    * Alanine aminotransferase/aspartate aminotransferase (ALT/AST) < 5 times the upper limit of the normality
    * Total bilirubin < 3 x institutional upper limit of normal (IULN)
    * Creatinine < 2.5 times the upper limit of the normality
    * Azithromycin allowed but if on both drugs patient should be on constant cardiovascular (CV) monitoring
    * Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessment/procedures being conducted
    * Subject is willing and able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Pleural effusion > grade 2 evident on chest x-ray (CXR) or chest computed tomography (CT)
* Intubation/mechanical ventilation
* Known hypersensitivity to dasatinib
* Patient being treated with immunomodulators or anti-rejection drugs
* Known active infections or other clinical condition that contraindicate dasatinib and cannot be treated or solved according to the judgement of the clinician
* ALT/AST > 5 times the upper limit of the normality
* Total bilirubin > 3 x IULN
* Neutrophils < 1000 / mmc unless; platelets < 50,000 / mmc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants requiring invasive mechanical ventilation, requiring tocilizumab or dying | Up to 28 days
  Outcome reported as the number of patients requiring mechanical ventilation, requiring tocilizumab or dying.

SECONDARY OUTCOMES:
Absolute lymphocyte count | Baseline, during treatment (day 1-14) up to 1 month
  Assessment via standard blood chemistry and metabolic panel
CRP (C-reactive protein) level | Baseline, during treatment (day 1-14) up to 1 month
  Assessment via standard blood chemistry and metabolic panel
Change of the SOFA (Sequential Organ Failure Assessment) | Baseline, during treatment (day 1-14) up to 1 month
  The SOFA score assessment will be based on PaO2/FiO2, platelets, Glasgow coma scale (GCS), bilirubin, Mean arterial pressure OR administration of vasoactive agents required, and Serum creatinine
Number of participants with treatment-related side effects | During treatment and up to 30 days after the last treatment dose
  Outcome reported as the number of adverse events and serious adverse events that occurred.
Radiological response | Baseline (optional), after seven days and if clinically indicated(up to 1 month)
  Will be evaluated by chest x-ray or pulmonary computed tomography (CT)
Duration of hospitalization | From baseline up to patient's discharge (up to 1 month)
  Outcome reported as the duration of hospitalization of patients
Remission of respiratory symptoms | Up to 1 month
  Time to invasive mechanical ventilation (if not previously initiated) calculated from baseline to intubation.
Remission of respiratory symptoms | Up to 1 month
  Time to definitive extubation calculated from intubation (any time occurred) to extubation in days.
Remission of respiratory symptoms | Up to 1 month
  Time to independence from oxygen therapy in days.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Mohrbacher, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States